CLINICAL TRIAL: NCT01041144
Title: Effects of Health Care Provider-mediated, Remote Coaching System Through the PDA-type Glucometer and the Internet on Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Ministry for Health Welfare and Family Affairs (Unknown)
Purpose: Supportive Care
Other Study IDs: Seoul R&D Project
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2009-12-31 (Estimated); Status verified 2005-06

CONDITIONS: Type 2 Diabetes; Lifestyle Intervention; Glucose Control; Internet Communication
Keywords: Diabetes; PDA; Internet; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: lifestyle counseling

INTERVENTIONS:
Behavioral: lifestyle counseling — supporting diabetes patients using Internet communication

SUMMARY:
The purpose of this study is to investigate the effectiveness of the new diabetes care delivery system applied to preexisting public health care resources through advanced information technologies such as PDA-type glucometer and the Internet on the glycemic control of type 2 diabetes patients lived in isolated rural area.

The investigators conducted a prospective, randomized, controlled trial in patients with type 2 diabetes for 12 weeks. The intervention group was treated with the new health care delivery system, where diabetes center provided specialized management, mediated by nurse of primary health care posts using the Internet and the PDA-type glucometer, while the control group with conventional health care. HbA1c, fasting plasma glucose and lipids levels were measured at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients
* Aged ≥ 40 years
* Baseline HbA1c of 7.0 to 11.0 % who had been already followed up for more than 6 months in the health care post

Exclusion Criteria:

* Participants with diagnosed or suspected disease of the liver, pancreas, endocrine organs, or kidney
* Ischemic heart disease or cerebrovascular disease or a history of such disease
* A creatinine level > 0.133 mmol/L
* Treatment with an intensified insulin regimens and those unable .

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 115

PRIMARY OUTCOMES:
HbA1c

SECONDARY OUTCOMES:
PP2hr Lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ho Yoon, Ph.D., Principal Investigator — Catholic Medical College
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea